CLINICAL TRIAL: NCT04345796
Title: Multicenter, Randomized, 2 x 2 Factorial, Phase 3 Study to Assess the Efficacy of Carvedilol and Empagliflozin on Improvement of Right Ventricular Remodeling in Patients With Severe Functional Tricuspid Regurgitation
Brief Title: Pharmacological Reduction of Right Ventricular Enlargement
Acronym: PROVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corporation (Unknown)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-0127
Record Dates: First submitted 2020-04-12; First posted 2020-04-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Tricuspid Regurgitation; Right Ventricular Dilatation
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — Carvedilol; empagliflozin

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial
Who Masked: Outcomes Assessor
Masking Description: To study efficacy of carvedilol, participants will be assigned to a carvedilol or to placebo and the identity of the treatment will be concealed by the use of study drugs that are identical in packaging, labeling, appearance and odor. Participants allocated to the SGLT2 inhibitor arm will receive empagliflozin 10mg.
  All imaging studies will be analyzed by core laboratory investigators who will be blinded to treatment assignment from the time of randomization until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- carvedilol+empagliflozin (Active Comparator): Patients will receive carvedilol SR 16mg and empagliflozin 10mg qd.
  Interventions: Drug: Carvedilol+Empagliflozin
- carvedilol alone (Active Comparator): Patients will receive carvedilol SR 16mg alone.
  Interventions: Drug: Carvedilol
- empagliflozin alone (Active Comparator): Patients will receive empagliflozin 10mg and matching placebo of carvedilol.
  Interventions: Drug: Empagliflozin
- placebo (Placebo Comparator): Patients will receive matching placebo of carvedilol.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol+Empagliflozin — Group A
  Other Names: Dilatrend SR+Jardiance
  Arms: carvedilol+empagliflozin
Drug: Carvedilol — Group B
  Other Names: Dilatrend SR
  Arms: carvedilol alone
Drug: Empagliflozin — Group C
  Other Names: Jardiance
  Arms: empagliflozin alone
Drug: Placebo — Group D
  Other Names: Matching placebo of Dilatrend SR
  Arms: placebo

SUMMARY:
Functional tricuspid regurgitation (TR) has been regarded as a secondary phenomenon of heart failure (HF), mitral valve (MV) disease or atrial fibrillation. Regardless of left ventricular (LV) function or pulmonary artery pressure, presence of moderate or greater functional TR is associated with poor prognosis. When a patient develops functional TR, it causes RV dilation and tricuspid annular enlargement, which also lead to deterioration of TR. A vicious cycle of significant TR, RV volume overload, tricuspid annular dilation and consequent aggravation of TR is accepted as a main determinant of the poor clinical outcome of patients with TR. Therefore, therapies that induce reverse remodeling of the RV and consequently reduce TR, may improve clinical outcomes. However, there have been no proven medical therapies for TR. The investigators hypothesize that carvedilol or empagliflozin is effective on improving RV remodeling in patients with functional severe TR and try to examine this hypothesis in a multicenter, 2x2 factorial, and randomized comparison study using cardiac MRI.

DETAILED DESCRIPTION:
Functional tricuspid regurgitation (TR) has been regarded as a secondary phenomenon of heart failure (HF), mitral valve (MV) disease or atrial fibrillation. The prevalence of functional TR was reported to be 25-64% in patients with either ischemic or non-ischemic cardiomyopathy. Regardless of left ventricular (LV) function or pulmonary artery pressure, presence of moderate or greater functional TR is associated with poor prognosis. When a patient develops functional TR, it causes RV dilation and tricuspid annular enlargement, which also lead to deterioration of TR. A vicious cycle of significant TR, RV volume overload, tricuspid annular dilation and consequent aggravation of TR is accepted as a main determinant of the poor clinical outcome of patients with TR. Because the quantitative assessment of RV size and function using echocardiography is often limited due to the complex geometry of RV, cardiac magnetic resonance imaging (MRI) has emerged as a gold standard for evaluating RV volume and function with excellent accuracy and reproducibility. The investigators previously reported that RV end-systolic volume index (ESVI) and RV end-diastolic volume index (EDVI) measured by MRI were significantly larger in severe TR patients, and also found that preoperative RV ESVI and RV ejection fraction (EF) on MRI were independent predictors of cardiac death and postoperative adverse events in patients who underwent TV surgery for severe functional TR. Therefore, therapies that induce reverse remodeling of the RV and consequently reduce TR, may improve clinical outcomes. However, there have been no proven medical therapies for TR. The morbidity and mortality of patients with functional TR remain high and novel therapeutic agents are needed to improve the prognosis of patients with functional TR. The investigators hypothesize that carvedilol or empagliflozin is effective on improving RV remodeling in patients with functional severe TR and try to examine this hypothesis in a multicenter, 2x2 factorial, and randomized comparison study using cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree to the study protocol and provide written informed consent
* Outpatients ≥ 20 years of age, male or female
* Patients with severe functional tricuspid regurgitation

  * TR whose vena contracta ≥0.7cm or central jet area > 10 square cm and which lasted > 6 months under medical treatment
  * LV ejection fraction ≥ 50%
* Dyspnea of NYHA functional class II or III

Exclusion Criteria:

* History of hypersensitivity or allergy to the study drugs, drugs of similar chemical classes, as well as known or suspected contraindications to the study drug
* Current use or prior use of a SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor
* Significant left-sided valve disease
* Left ventricular ejection fraction <40%
* Marked bradycardia (<50 beats/min) or 2nd or 3rd degree AVB, sinus node dysfunction
* Severe pulmonary hypertension: TR Vmax >4m/s at screening (including Cor pulmonale)
* Medical history of hospitalization within 6 weeks
* Current acute decompensated heart failure or dyspnea of NYHA functional class IV
* Symptomatic hypotension and/or a SBP < 90 mmHg at screening Estimated GFR < 30 mL/min/1.73 square m
* History of ketoacidosis, Type 1 diabetes
* Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 2 x upper limit of normal (ULN) at screening visit (Visit 0), history of hepatic encephalopathy, history of esophageal varices, or history of portocaval shunt.
* Acute coronary syndrome, stroke, severe peripheral artery disease or major CV surgery or PCI within 3 months
* History of severe pulmonary disease (asthma, COPD with bronchial hypersensitivity)
* Secondary hypertension such as pheochromocyotoma
* Acute pulmonary thromboembolism
* Variant angina, vocal cord edema, severe allergic rhinitis
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using a barrier method plus a hormonal method
* Pregnant or nursing (lactating) women
* Contraindication for MRI

  * Presence of pacemaker or ICD, implanted metallic objects, claustrophobia
  * Severe beat-to-beat variation
* Galactose intolerance, Lapp lactose deficiency, glucose-galactose malabsorption
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Change of RV end-systolic volume index | from baseline to 12 months follow-up
  Change of RV end-systolic volume index by cardiac MRI

SECONDARY OUTCOMES:
Change of RV end-diastolic volume index | from baseline to 12 months follow-up
  Change of RV end-diastolic volume index by cardiac MRI
Change of RV ejection fraction | from baseline to 12 months follow-up
  Change of RV ejection fraction by cardiac MRI
Change of vena contract width of TR | from baseline to 12 months follow-up
  Change of vena contract width of TR by echocardiography
Occurrences of death from cardiovascular causes or hospitalization for heart failure | the entire follow-up period (continuing until 12 months after the last patient was enrolled)
  Clinical outcome
Occurrences of death from any causes | the entire follow-up period (continuing until 12 months after the last patient was enrolled)
  Clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: DUK HYUN KANG, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided